CLINICAL TRIAL: NCT04454125
Title: Air Quality Index (AQI) and Childhood Asthma: an Intervention
Brief Title: AQI and Childhood Asthma: an Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: American Thoracic Society (Other)
Responsible Party: Principal Investigator, Franziska Rosser, MD MPH, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19120083
Record Dates: First submitted 2020-06-26; First posted 2020-07-01 (Actual); Results first posted 2023-08-15 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Asthma; Asthma in Children
Keywords: Air Quality Index (AQI); Childhood asthma exacerbations
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: 40 child will be 1:1 randomization by age groups 8-12 years, 13-17 years.
Masking Description: Unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (Active Comparator)
  Interventions: Other: Routine care
- AQI Intervention (Experimental)
  Interventions: Behavioral: AQI intervention

INTERVENTIONS:
Behavioral: AQI intervention — The intervention arm will receive AQI education, an asthma action plan containing AQI information and recommendations, and will be required to demonstrate ability to check AQI (either via airnow.gov website or downloaded AirNow smartphone app).
  Arms: AQI Intervention
Other: Routine care — The routine care arm will be provided with general AQI education and an asthma action plan not containing AQI information.
  Arms: Routine Care

SUMMARY:
This is a small pilot prospective intervention trial in children with asthma who will be randomized to receive either (A) Air Quality Index (AQI) education + an asthma action plan (control) or (B) AQI education + an asthma action plan which contains AQI behavioral recommendations + demonstrate ability to navigate to AirNow either online or on smartphone app (intervention).

DETAILED DESCRIPTION:
Over 3 million US children with asthma reported at least one attack in the prior year. Poorly controlled asthma is a major cause of suffering, school absences, loss of caregiver productivity, and healthcare costs (estimated as ~$80 billion/year). Over half of children on controller medication are not well controlled, due to environmental exposures, non-adherence, or true non-response to treatment. Outdoor air pollution is a known trigger of asthma. Although sound health policies are the best long-term approaches to reduce the harmful effects of air pollution, exposure avoidance is needed until "clean air" is ensured through effective legislation. Despite this, healthcare providers infrequently provide pollution exposure advice to children with asthma. The Environmental Protection Agency (EPA) monitors air pollution and reports a daily Air Quality Index (AQI) that is easy to use and available in most metropolitan areas. Practical recommendations regarding outdoor activity can be based on AQI levels. Despite this, AQI-based recommendations are rarely addressed in asthma action plans (AAP). No pediatric study has assessed the addition of the AQI to AAP to reduce asthma morbidity. This proposal seeks to recruit a pilot cohort of 40 children with asthma. Using this cohort, the investigators will test the hypotheses that (1) the addition of the AQI to AAP will reduce asthma exacerbations and (2) the addition of the AQI to AAP will improve asthma symptom control & quality of life in children with asthma. The inclusion of the AQI onto asthma action plans is novel in clinical asthma care; its wide availability would make large-scale implementation feasible. The investigators expect this low-cost and low-tech intervention will have a positive impact in reducing asthma morbidity. Given that 1 out of every 12 children in the U.S. has asthma, this is relevant to health care professionals, parents, and public health practitioners.

Optional, the investigators will collect nasal epithelial cells for use in future genomic/epigenetic studies.

Additionally, 40 parents/guardians of the children were also recruited to complete a baseline parental knowledge and usage of the AQI questionnaire administered at the randomization visit. This was originally listed as a secondary outcome however was removed during reporting of results as parental knowledge is not a true clinical trial outcome. Also, the secondary outcome of baseline child AQI usage (checking AQI) was changed to reflect this was a measure collected at all study visits and the secondary measure of physical activity was added.

ELIGIBILITY:
Inclusion Criteria:

* Child Inclusion criteria includes:

  1. physician diagnosis of persistent asthma- either mild, moderate, or severe;
  2. family home internet access and/or smartphone access + willingness to download AirNow app on phone;
  3. age 8-17 years.

Parent/guardian inclusion: parent or guardian of the child participant, of whom has met inclusion criteria.

Exclusion Criteria:

* Child exclusion criteria includes:

  1. diagnosis of other chronic respiratory disease (e.g. cystic fibrosis, bronchopulmonary dysplasia, etc)
  2. immunodeficiency- acquired or congenital
  3. neuromuscular disease
  4. disability affecting ambulation
  5. cyanotic congenital heart disease
  6. only 1 child per household eligible
  7. no plans to leave Pittsburgh area in next 6 months

Parental/guardian exclusion criteria: none.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2021-03-22 (Actual); Study Completion 2021-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Rosser, MD MPH, Principal Investigator — UPMC | Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not currently have an individual participant data sharing plan. However, de-identified research data/documents may be shared in the future with other investigators who share similar research interests.
  Specimens and data will not be released without (1) PI written permission and (2) appropriate Institutional Review Board (IRB) approval. Data use and/or material transfer agreements will also be required as applicable to outside researchers.

REFERENCES:
- [Background] Reyes-Angel J, Han YY, Forno E, Celedon JC, Rosser FJ. Parental knowledge and usage of air quality in childhood asthma management. Front Pediatr. 2022 Oct 26;10:966372. doi: 10.3389/fped.2022.966372. eCollection 2022. PMID 36440347
- [Result] Rosser FJ, Rothenberger SD, Han YY, Forno E, Celedon JC. Air Quality Index and Childhood Asthma: A Pilot Randomized Clinical Trial Intervention. Am J Prev Med. 2023 Jun;64(6):893-897. doi: 10.1016/j.amepre.2022.12.010. Epub 2023 Jan 13. PMID 36642643

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Care | AQI Intervention
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care | AQI Intervention | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 20 | 40
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.5 (2.6) | 12.5 (2.9) | 12.5 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9 | 6 | 15
  More than 1 race | 3 | 4 | 7
  White | 8 | 10 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 20 | 40
At least one severe asthma exacerbation in the past 12 months, yes [Count of Participants; unit: Participants] | 11 | 13 | 24
Asthma Control Test (ACT) [Mean (Standard Deviation); unit: score on a scale] — ACT score ranges from 5-25. Scores <=19 concerning for poor asthma control, scores <=15 concerning for very poor asthma control Population: ACT administered to children aged 12 years and older.
  score on a scale
    number analyzed (Participants) | 13 | 13 | 26
    (all) | 20.9 (4.6) | 21.2 (3.0) | 21.0 (3.8)
Childhood Asthma Control Test (CACT) [Mean (Standard Deviation); unit: score on a scale] — CACT score ranges from 0-27. Scores <=19 concerning for poor asthma control, scores <=12 concerning for very poor asthma control Population: CACT administered to children aged 8-11 years of age
  score on a scale
    number analyzed (Participants) | 7 | 7 | 14
    (all) | 22.6 (1.3) | 20.7 (8.3) | 21.6 (5.8)
Pediatric Asthma Quality of Life Questionnaire [Mean (Standard Deviation); unit: score on a scale] — PAQLQ scores range from 1 (severe asthma impairment) to 7 (no asthma impairment)
  score on a scale | 5.96 (1.02) | 6.11 (0.84) | 6.03 (0.93)
Body Mass Index z-score (BMIz) [Mean (Standard Deviation); unit: z score] — BMI is calculated by dividing a child's weight (in kg) by height squared (in meters), age and sex specific, and expressed as z-scores which are based on standard normal distribution. A score of 0 represents the population mean. For children, a BMI z-score equal to or greater than 1.036 and less than 1.645 is defined as overweight. A z-score equal to or greater than 1.645 is defined as obese. Reference: Center for Disease Control and Prevention (CDC) growth charts.
  z score | 1.51 (1.35) | 1.03 (1.22) | 1.27 (1.29)
Reported checking the AQI prior to going outside to be active, yes [Count of Participants; unit: Participants] | 2 | 2 | 4
Reported any change in outdoor activity because of the AQI, yes [Count of Participants; unit: Participants] | 5 | 3 | 8
Reported moderate or vigorous activity for at least 10 minutes outside in a typical week, yes [Count of Participants; unit: Participants] | 14 | 18 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Moderate or Severe Asthma Exacerbation Over Time
Description: Moderate and severe asthma exacerbations were captured via questionnaire administered monthly for up to 6 months. Severe and moderate exacerbations were defined by American Thoracic Society (ATS) criteria.
Time Frame: Over study duration (up to 6 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | AQI Intervention
Number analyzed (Participants) | 20 | 20
Participants
  At least one severe asthma exacerbation during study, yes | 5 | 4
  At least one moderate asthma exacerbation during study, yes | 13 | 12
Statistical Analysis 1: Comparison: Routine Care vs AQI Intervention; Outcome= severe asthma exacerbation at visit (yes, no), collected via questionnaire at visits 2-7(exit). Does not include randomization (visit 1); Test type: Superiority; p = 0.32, Generalized linear model, repeat measure; Generalized linear model (GLM) fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.23 to 1.61] — Estimate is for the control group (Routine Care) obtained from generalized linear model with repeat measures including group arm, visit, interaction term (arm*visit) and adjusting for visit 2 severe asthma exacerbation
Statistical Analysis 2: Comparison: Routine Care vs AQI Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.29, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.03 to 2.76] — Estimate is for the intervention group (AQI intervention) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit) and adjusting for visit 2 severe asthma exacerbation
Statistical Analysis 3: Comparison: Routine Care vs AQI Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.58, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.51, 95% CI 2-sided [0.05 to 5.68]; Estimate is for the interaction term (group*visit) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit) and adjusting for visit 2 severe asthma exacerbation
Statistical Analysis 4: Comparison: Routine Care vs AQI Intervention; Outcome= moderate asthma exacerbation at visit (yes, no), collected via questionnaire at visits 2-7(exit). Does not include randomization (visit 1); Test type: Superiority; p = 0.02, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.50, 95% CI 2-sided [0.27 to 0.91] — Estimate is for the control group (Routine Care) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit) and adjusting for visit 2 moderate asthma exacerbation
Statistical Analysis 5: Comparison: Routine Care vs AQI Intervention; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.03, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.23, 95% CI 2-sided [0.06 to 0.86] — Estimate is for the intervention group (AQI Intervention) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit) and adjusting for visit 2 moderate asthma exacerbation
Statistical Analysis 6: Comparison: Routine Care vs AQI Intervention; [analysis description as in outcome 1, analysis 4]; Test type: Superiority; p = 0.30, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.11 to 1.95] — Estimate is for the interaction term (group*visit) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit) and adjusting for visit 2 moderate asthma exacerbation

2. Primary Outcome: Mean Change in Asthma Control Over Time
Description: Asthma symptom control was measured by the validated Asthma Control Test (ACT) or Childhood Asthma Control Test (CACT) questionnaires as age appropriate (ACT in children 12 year of age or older; CACT for children younger than 12 years of age). ACT and CACT were obtained at baseline and every 4 weeks for up to 6 months. Differences in asthma control scores were compared both within arms and between arms at study end. ACT (min=5, max=25, score of <=19 concerning for poor asthma control; <=15 concerning for very poorly controlled). CACT (min=0, max=27, score of <=19 concerning for poor asthma control; <=12 concerning for very poorly controlled)
Time Frame: Over study duration (up to 6 months)
Population: The mean change was obtained, via generalized linear modeling (glm), taking into account the correlation of repeat measures. The values are listed by group and contain all available time points averaged.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Routine Care | AQI Intervention
Number analyzed (Participants) | 20 | 20
score on a scale
  Asthma Control Test: number analyzed (Participants) | 13 | 13
  Asthma Control Test | 0.17 [-1.17 to 1.51] | 2.02 [0.88 to 3.15]
  Childhood Asthma Control Test: number analyzed (Participants) | 7 | 7
  Childhood Asthma Control Test | -0.31 [-1.87 to 1.25] | 3.96 [-1.27 to 9.20]
Statistical Analysis 1: Comparison: Routine Care vs AQI Intervention; Outcome=Asthma Control Test Score. Obtained at all visits; Test type: Superiority; p = 0.80, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 0.17, 95% CI 2-sided [-1.17 to 1.51] — Estimate is for the control group (Routine Care) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit)
Statistical Analysis 2: Comparison: Routine Care vs AQI Intervention; Outcome=Asthma Control Test Score. Obtained at all visits; Test type: Superiority; p = 0.001, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 2.02, 95% CI 2-sided [0.88 to 3.15] — Estimate is for the intervention group (AQI Intervention) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit)
Statistical Analysis 3: Comparison: Routine Care vs AQI Intervention; Outcome=Asthma Control Test Score. Obtained at all visits; Test type: Superiority; p = 0.04, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 1.85, 95% CI 2-sided [0.09 to 3.61] — Estimate is for the interaction term (group*visit) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit)
Statistical Analysis 4: Comparison: Routine Care vs AQI Intervention; Outcome=Childhood Asthma Control Test Score. Obtained at all visits; Test type: Superiority; p = 0.70, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = -0.31, 95% CI 2-sided [-1.87 to 1.25] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Routine Care vs AQI Intervention; Outcome=Childhood Asthma Control Test Score. Obtained at all visits; Test type: Superiority; p = 0.14, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 3.96, 95% CI 2-sided [-1.27 to 9.20] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 6: Comparison: Routine Care vs AQI Intervention; Outcome=Childhood Asthma Control Test Scores; Test type: Superiority; p = 0.13, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 4.27, 95% CI 2-sided [-1.19 to 9.73] — [estimate comment as in outcome 2, analysis 3]

3. Primary Outcome: Mean Change in Pediatric Asthma Quality of Life Over Time
Description: Quality of life will be measured by the validated Pediatric Asthma Quality of Life Questionnaire with standardized activities (PAQLQ) at entrance and exit visits. Differences in PAQLQ scores will be compared both within arms and between arms at study end. PAQLQ (min=1 (extremely bothered/all the time), max=7 (not bothered/none of the time)
Time Frame: Baseline, 6 months
Population: 1 participant lost to follow up at exit visit
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Routine Care | AQI Intervention
Number analyzed (Participants) | 20 | 19
score on a scale | 0.25 [-0.06 to 0.55] | 0.54 [0.20 to 0.88]
Statistical Analysis 1: Comparison: Routine Care vs AQI Intervention; Outcome: Pediatric Asthma Quality of Life Questionnaire. Obtained at randomization and exit visits (visit 1 and visit 7); Test type: Superiority; p = 0.11, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 0.25, 95% CI 2-sided [-0.06 to 0.55] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Routine Care vs AQI Intervention; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.002, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 0.54, 95% CI 2-sided [0.20 to 0.88] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Routine Care vs AQI Intervention; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.20, generalized linear model, repeat measure; GLM fitted with Normal/Gaussian distribution and identity link; Mean Difference (Net) = 0.30, 95% CI 2-sided [-0.16 to 0.75] — [estimate comment as in outcome 2, analysis 3]

4. Secondary Outcome: Number of Participants Who Reported Checking the AQI Prior to Going Outside to be Active
Description: Participant reported checking of AQI prior to going outside to be active assessed via questionnaire. Question: In the past 4 weeks, did you check the air quality index before going outside to be active? Response choices: Yes, No.
Time Frame: Over study duration, assessed at baseline and monthly during study for up to 6 months. Reported below at exit.
Population: 1 participant lost to follow up at exit visit; all participant data (n=40) was included in glm analyses as presented in statistical analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | AQI Intervention
Number analyzed (Participants) | 20 | 19
Participants | 3 | 12
Statistical Analysis 1: Comparison: Routine Care vs AQI Intervention; Outcome: Reported checking the AQI prior to going outside to be active; Test type: Superiority; p = 0.87, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.45 to 1.96] — Estimate is control group (Routine Care) obtained from generalized linear model with repeat measures including group, visit, interaction term (group*visit)
Statistical Analysis 2: Comparison: Routine Care vs AQI Intervention; Outcome: Reported checking the AQI prior to going outside to be active; Test type: Superiority; p = 0.004, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 6.89, 95% CI 2-sided [1.85 to 25.6] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Routine Care vs AQI Intervention; Outcome: Reported checking the AQI prior to going outside to be active; Test type: Superiority; p = 0.01, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 7.31, 95% CI 2-sided [1.62 to 32.9] — [estimate comment as in outcome 2, analysis 3]

5. Secondary Outcome: Number of Participated Who Reported Outdoor Activity Behavioral Change in Response to the AQI
Description: Usage of the AQI prior to exercise was monitored monthly via questionnaire. Question: In the past 4 weeks, how many times did you change your outdoor activity because of the air quality index? Response choices: All of the time, Most of the time, Some of the time, A little of the time, None of the time. A positive response was considered an answer of all, most, some, or a little of the time. A negative response was considered none of the time.
Time Frame: Over study duration, assessed at baseline and monthly during study for up to 6 months. Reported below at exit.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | AQI Intervention
Number analyzed (Participants) | 20 | 19
Participants | 2 | 7
Statistical Analysis 1: Comparison: Routine Care vs AQI Intervention; Outcome: Reported outdoor activity behavioral change in response to the AQI, obtained at all visits; Test type: Superiority; p = 0.15, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.08 to 1.47] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Routine Care vs AQI Intervention; Outcome: Reported outdoor activity behavioral change in response to the AQI, obtained at all visits; Test type: Superiority; p = 0.94, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.35 to 2.68] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Routine Care vs AQI Intervention; Outcome: Reported outdoor activity behavioral change in response to the AQI, obtained at all visits; Test type: Superiority; p = 0.26, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 2.79, 95% CI 2-sided [0.47 to 16.5] — [estimate comment as in outcome 2, analysis 3]

6. Secondary Outcome: Number of Participants Who Reported Moderate or Vigorous Physical Activity for at Least 10 Minutes Continuously Outside in a Typical Week
Description: Outcome obtained from physical activity questionnaire. Yes represents a positive response to at least one of the follow two questions: Question 1: In a typical week {do you/does SP} do any vigorous-intensity sports, fitness, or recreational activities that cause large increases in breathing or heart rate like running or basketball for at least 10 minutes continuously outside? Response choices: Yes, No, Refused, Don't Know. Note: refused and don't know were coded as negative. Question 2: In a typical week, {do you/does SP} do any moderate-intensity sports, fitness, or recreational activities that cause a small increase in breathing or heart rate such as brisk walking, bicycling, swimming, or volleyball for at least 10 minutes continuously outside? Response choices: Yes, No, Refused, Don't Know. Note: refused and don't know were coded as negative.
Time Frame: Over study duration, assessed at baseline and monthly during study for up to 6 months. Reported below at exit.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | AQI Intervention
Number analyzed (Participants) | 20 | 19
Participants | 9 | 7
Statistical Analysis 1: Comparison: Routine Care vs AQI Intervention; Obtained at all visits; Test type: Superiority; p = 0.004, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.42, 95% CI 2-sided [0.24 to 0.76] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Routine Care vs AQI Intervention; Obtained at all visits; Test type: Superiority; p < 0.0001, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.05 to 0.31] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: Routine Care vs AQI Intervention; Obtained at all visits; Test type: Superiority; p = 0.03, generalized linear model, repeat measure; GLM fitted with binomial distribution and logit link; Odds Ratio (OR) = 0.29, 95% CI 2-sided [0.10 to 0.87] — [estimate comment as in outcome 2, analysis 3]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the 6 month study duration.
Description: Asthma is a chronic lung disease with varying impairment and risk, thus asthma exacerbations and loss of control are not unexpected. However, if a participant reported 3 severe asthma exacerbations, 3 consecutive control test scores <=19, or had FEV1 <80% at either visit, these were recorded, the parent was notified, and follow-up with managing asthma specialist was recommended. Hospitalizations for asthma were considered expected, serious adverse events.
Arm/Group | Routine Care | AQI Intervention
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/20
Other Adverse Events (participants affected / at risk) | 3/20 | 4/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Care (N=20) | AQI Intervention (N=20)
Asthma exacerbation requiring hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Routine Care (N=20) | AQI Intervention (N=20)
Three consecutive poor control scores (Respiratory, thoracic and mediastinal disorders) | 3 | 1 — Having 3 consecutive ACT or CACT scores concerning for poor control (<=19)
Three severe asthma exacerbations (Respiratory, thoracic and mediastinal disorders) | 2 | 0 — Reporting a severe asthma exacerbation at 3 study visits
Low FEV1 (Respiratory, thoracic and mediastinal disorders) | 2 | 3 — Forced expiratory volume in 1 sec (FEV1) <80% at randomization or exit visit

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04454125/Prot_SAP_000.pdf